CLINICAL TRIAL: NCT01245751
Title: Safety, Tolerability and Immunogenicity of a Booster Dose of ZOSTAVAX™ Administered ≥10 Years After a First Dose Compared With a First Dose of ZOSTAVAX™
Brief Title: Safety, Tolerability, and Immunogenicity of a Booster Dose of Zoster Vaccine, Live (V211-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: University of Colorado, Denver (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V211-029
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster; Varicella-zoster Vaccine
Keywords: Shingles; Vaccine
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Booster Dose Participants ≥70 years of age (Experimental): Herpes zoster history-negative participants ≥70 years of age who received Zoster Vaccine, Live approximately 10 years prior in the Shingles Prevention Study V211-004 NCT00007501)
  Interventions: Biological: Zoster Vaccine, Live
- Group 2: First Dose Participants ≥70 years of age (Experimental): Herpes zoster history-negative participants ≥70 years of age who have never received Zoster Vaccine, Live and are matched to Group 1 participants by age
  Interventions: Biological: Zoster Vaccine, Live
- Group 3: First Dose Participants ≥60 and <70 years of age (Experimental): Herpes zoster history-negative participants ≥60 and <70 years of age who have never received Zoster Vaccine, Live
  Interventions: Biological: Zoster Vaccine, Live
- Group 4: First Dose Participants ≥50 and <60 years of age (Experimental): Herpes zoster history-negative participants ≥50 and <60 years of age who have never received Zoster Vaccine, Live
  Interventions: Biological: Zoster Vaccine, Live

INTERVENTIONS:
Biological: Zoster Vaccine, Live — Single approximately 0.65-mL subcutaneous injection of Zoster Vaccine, Live on Day 1 of the study
  Other Names: V211; ZOSTAVAX™

SUMMARY:
This study was conducted to obtain safety and immunogenicity data after a booster dose of Zoster Vaccine, Live administered ≥10 years following an initial dose. This information was compared to similar information obtained after Zoster Vaccine, Live administration to age-matched and younger participants who received their first dose of Zoster Vaccine, Live. The study was designed to determine: 1) whether a booster dose of Zoster Vaccine, Live in participants ≥70 years of age induces an antibody response that is noninferior to that of a first dose of Zoster Vaccine, Live in participants matched for age; 2) whether a booster dose of Zoster Vaccine, Live induces an acceptable rise in the level of varicella-zoster virus (VZV) antibodies.

DETAILED DESCRIPTION:
All participants were followed for one year after completion of the 42-day post-vaccination period while Groups 1 and 2 were followed for a total of three years.

ELIGIBILITY:
Inclusion Criteria:

* All Groups:

  * Must not have a fever of ≥100.4° F on the day of vaccination
  * Any underlying chronic illness must be in stable condition
  * History of varicella or residence in a VZV-endemic area for ≥30 years
* Group 1:

  * 70 years of age or older
  * Took part in the Shingles Prevention Study (SPS) (V211-004, NCT00007501) and received a single dose of Zoster Vaccine, Live ≥10 years prior to enrollment in this study
* Group 2:

  * 70 years of age or older
* Group 3:

  * 60 to 69 years of age
* Group 4:

  * 50 to 59 years of age

Exclusion Criteria:

* All Groups:

  * History of hypersensitivity reaction to any vaccine component or an anaphylactic/anaphylactoid reaction to neomycin
  * Prior history of herpes zoster
  * Pregnant or breast-feeding, or expecting to conceive within the duration of the study
  * Has been treated with immunoglobulin or any blood products, other than autologous (self-donated) blood transfusion, in the 5 months prior to vaccination
  * Received any other vaccine within 4 weeks prevaccination
  * On immunosuppressive therapy
  * Has known or suspected immune dysfunction
  * Is taking any non-topical antiviral therapy with activity against herpesviruses, including, but not limited to acyclovir, famciclovir, valacyclovir, and ganciclovir.
* Groups 2, 3, and 4:

  * Has previously received any varicella or zoster vaccine

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Levin MJ, Schmader KE, Pang L, Williams-Diaz A, Zerbe G, Canniff J, Johnson MJ, Caldas Y, Cho A, Lang N, Su SC, Parrino J, Popmihajlov Z, Weinberg A. Cellular and Humoral Responses to a Second Dose of Herpes Zoster Vaccine Administered 10 Years After the First Dose Among Older Adults. J Infect Dis. 2016 Jan 1;213(1):14-22. doi: 10.1093/infdis/jiv480. Epub 2015 Oct 9. PMID 26452397
- [Derived] Weinberg A, Popmihajlov Z, Schmader KE, Johnson MJ, Caldas Y, Salazar AT, Canniff J, McCarson BJ, Martin J, Pang L, Levin MJ. Persistence of Varicella-Zoster Virus Cell-Mediated Immunity After the Administration of a Second Dose of Live Herpes Zoster Vaccine. J Infect Dis. 2019 Jan 7;219(2):335-338. doi: 10.1093/infdis/jiy514. PMID 30165651

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Booster Dose Participants ≥70 Years of Age: Herpes zoster history-negative participants ≥70 years of age who received Zoster Vaccine, Live approximately 10 years prior in the Shingles Prevention Study V211-004 (NCT00007501). Participants received a single Zoster Vaccine, Live vaccination on Day 1.
- Group 2: First Dose Participants ≥70 Years of Age: Herpes zoster history-negative participants ≥70 years of age who have never received Zoster Vaccine, Live and are matched to Group 1 participants by age. Participants received a single Zoster Vaccine, Live vaccination on Day 1.
- Group 3: First Dose Participants ≥60 and <70 Years of Age: Herpes zoster history-negative participants ≥60 and <70 years of age who have never received Zoster Vaccine, Live. Participants received a single Zoster Vaccine, Live vaccination on Day 1.
- Group 4: First Dose Participants ≥50 and <60 Years of Age: Herpes zoster history-negative participants ≥50 and <60 years of age who have never received Zoster Vaccine, Live. Participants received a single Zoster Vaccine, Live vaccination on Day 1.
Period: Part 1: Day 1 to Week 52 (1 Year)
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age | Group 3: First Dose Participants ≥60 and <70 Years of Age | Group 4: First Dose Participants ≥50 and <60 Years of Age
Started | 201 | 199 | 100 | 100
Completed 42-day Postvaccination Period | 201 | 199 | 100 | 100
Completed | 199 | 194 | 100 | 98
Not Completed | 2 | 5 | 0 | 2
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 0 | 0
Period: Part 2: Week 156 (3 Year) Visit
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age | Group 3: First Dose Participants ≥60 and <70 Years of Age | Group 4: First Dose Participants ≥50 and <60 Years of Age
Started | 161 (Enrollment in Part 2 was voluntary) | 139 (Enrollment in Part 2 was voluntary) | 0 (Part 2 was planned for Groups 1 and 2 only) | 0 (Part 2 was planned for Groups 1 and 2 only)
Completed | 161 | 139 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age | Group 3: First Dose Participants ≥60 and <70 Years of Age | Group 4: First Dose Participants ≥50 and <60 Years of Age | Total
Number analyzed (Participants) | 201 | 199 | 100 | 100 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.1 (4.5) | 76.3 (5.1) | 64.1 (3.1) | 55.5 (2.8) | 71.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 94 | 65 | 77 | 343
  Male | 94 | 105 | 35 | 23 | 257

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of the Antibody Responses to Varicella-Zoster Virus (VZV)
Description: VZV antibody titers were determined by glycoprotein enzyme-linked immunosorbent assay (gpELISA)
Time Frame: Day 1 (Baseline) and Week 6 postvaccination
Population: Analysis included all vaccinated participants except those who had protocol deviations that interfered with the assessment of VZV antibody response, who developed varicella or herpes zoster rashes before a blood sample was taken, or who reported exposure to varicella or herpes zoster. The planned analysis included Group 1 versus Group 2 only.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA Units/mL
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age
Number analyzed (Participants) | 201 | 199
gpELISA Units/mL
  Day 1 (Baseline), n=201, 199 | 248.0 [219.7 to 280.0] | 254.2 [223.5 to 289.3]
  Week 6 postvaccination, n=198, 195 | 389.1 [351.4 to 430.8] | 368.6 [330.5 to 411.6]
Statistical Analysis 1: Comparison: Group 1: Booster Dose Participants ≥70 Years of Age vs Group 2: First Dose Participants ≥70 Years of Age; Week 6 analysis; Test type: Non-Inferiority or Equivalence — Week 6 GMT value for Group 1 is statistically non-inferior to Group 2 for the prespecified clinically relevant 1.5-fold ratio if the lower bound of the 95% confidence interval for the GMT ratio is >0.67; p < 0.001, Longitudinal regression model — The alpha threshold for statistical significance is 0.025 (1-sided); The analyzed GMT ratio, 95% confidence interval, and P-value were based on a longitudinal regression model adjusting for age and vaccination group; GMT Ratio = 1.05, 95% CI 2-sided [0.97 to 1.15]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) From Day 1 (Baseline) to Week 6 Postvaccination in VZV Antibody Titers
Description: VZV antibody titers were determined by gpELISA. The GMFR measures the rise in VZV antibodies from Day 1 (Baseline) to Week 6 postvaccination.
Time Frame: Day 1 (Baseline) and Week 6 postvaccination
Population: Analysis included all vaccinated participants except those who had protocol deviations that interfered with the assessment of VZV antibody response, who developed varicella or herpes zoster rashes before a blood sample was taken, or who reported exposure to varicella or herpes zoster. The planned analysis included Group 1 only.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Groups:
- Group 1: Booster Dose Participants ≥70 Years of Age: Herpes zoster history-negative participants ≥70 years of age who received Zoster Vaccine, Live approximately 10 years prior in the Shingles Prevention Study V211-004(NCT00007501). Participants received a single Zoster Vaccine, Live vaccination on Day 1.
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age
Number analyzed (Participants) | 198
Fold Rise | 1.5 [1.4 to 1.6]
Statistical Analysis 1: Comparison: Group 1: Booster Dose Participants ≥70 Years of Age; A booster dose induces a statistically acceptable VZV antibody response if the lower bound of the 95% confidence interval is >1.0; Test type: Superiority or Other; p < 0.001, Longitudinal regression model — The alpha threshold for statistical significance is 0.025 (1-sided); The analyzed GMFR, 95% confidence interval, and P-value were based on a longitudinal regression model adjusting for age; Geometric mean fold rise = 1.54, 95% CI 2-sided [1.44 to 1.66]

3. Secondary Outcome: Number of Participants Reporting One or More Adverse Experiences
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience. A serious adverse experience is any AE that results in death, is life threatening, results in persistent disability/incapacity, results in or prolongs existing inpatient hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is another important medical event that may jeopardize the participant and may require medical or surgical intervention. Vaccine-related AEs were those assessed by the investigator as definitely, probably, or possibly related to vaccine administration. This outcome measure applies only to AEs collected after vaccination in Part 1 of the current study.
Time Frame: Up to 42 days postvaccination
Population: Analysis included all vaccinated participants who had any safety follow-up
Measure: Number; unit: Participants
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age | Group 3: First Dose Participants ≥60 and <70 Years of Age | Group 4: First Dose Participants ≥50 and <60 Years of Age
Number analyzed (Participants) | 201 | 199 | 100 | 100
Participants
  Any Adverse Event | 104 | 95 | 72 | 72
  Injection-site Adverse Event | 68 | 61 | 56 | 57
  Non-Injection-site Adverse Event | 66 | 57 | 34 | 38
  Serious Adverse Event | 3 | 5 | 1 | 0
  Vaccine-related Serious Adverse Event | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days postvaccination: all AEs; Day 43 to Week 52: SAEs only; Week 156: SAEs only within 24 hours of the Week-156 blood draw (Groups 1 and 2 only)
Arm/Group | Group 1: Booster Dose Participants ≥70 Years of Age | Group 2: First Dose Participants ≥70 Years of Age | Group 3: First Dose Participants ≥60 and <70 Years of Age | Group 4: First Dose Participants ≥50 and <60 Years of Age
Serious Adverse Events (participants affected / at risk) | 29/201 | 29/199 | 6/100 | 2/100
Other Adverse Events (participants affected / at risk) | 76/201 | 58/199 | 61/100 | 62/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Booster Dose Participants ≥70 Years of Age (N=201) | Group 2: First Dose Participants ≥70 Years of Age (N=199) | Group 3: First Dose Participants ≥60 and <70 Years of Age (N=100) | Group 4: First Dose Participants ≥50 and <60 Years of Age (N=100)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Booster Dose Participants ≥70 Years of Age (N=201) | Group 2: First Dose Participants ≥70 Years of Age (N=199) | Group 3: First Dose Participants ≥60 and <70 Years of Age (N=100) | Group 4: First Dose Participants ≥50 and <60 Years of Age (N=100)
Injection-site erythema (General disorders) | 44 (44) | 47 (47) | 41 (41) | 40 (40)
Injection-site pain (General disorders) | 47 (47) | 28 (29) | 42 (46) | 48 (48)
Injection-site pruritus (General disorders) | 10 (10) | 9 (9) | 9 (9) | 11 (11)
Injection-site swelling (General disorders) | 31 (31) | 24 (24) | 29 (29) | 33 (33)
Nasopharyngitis (Infections and infestations) | 11 (11) | 2 (2) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 8 (11) | 4 (8) | 3 (3) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.